CLINICAL TRIAL: NCT00022568
Title: A Phase I Trial of Intra Lesional rV-Tricom Vaccine in the Treatment of Malignant Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068831; CPMC-IRB-14387; AECM-01-003; NCI-3353
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2003-12

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — rV-Tricom

INTERVENTIONS:
Biological: recombinant vaccinia-TRICOM vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of recombinant vaccinia-TRICOM vaccine in patients with metastatic melanoma.
* Determine the clinical toxic effects of this vaccine in these patients.
* Determine the safety of this vaccine in these patients.
* Determine the clinical response of these patients to this vaccine.
* Determine evidence of host anti-melanoma immune reactivity in these patients after treatment with this vaccine.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant vaccinia-TRICOM vaccine once every 4 weeks for a total of 3 vaccinations. Patients with stable or responding disease may receive an additional course of vaccinations.

Cohorts of 3-6 patients receive escalating doses of recombinant vaccinia-TRICOM vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline, at each vaccine administration, and at study completion.

Patients are followed at 3 months.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic non-resectable cutaneous, subcutaneous, or lymph node malignant melanoma
* Lesion(s) must be accessible to percutaneous injection
* Measurable lesion(s)

  * At least 1.0 cm
* Previously treated brain metastases with no evidence of disease or edema on MRI or CT scan allowed

  * At least 6 weeks since prior definitive therapy (surgery or radiotherapy)
* No untreated or edematous metastatic brain lesions or leptomeningeal disease
* No ascites or pleural effusions

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3
* Absolute granulocyte count at least 3,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic:

* Direct bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* No severe coagulation disorder with PT/PTT greater than 2 times normal (without anticoagulation medications)
* No hepatic insufficiency
* No alcoholic cirrhosis

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No renal insufficiency

Cardiovascular:

* No congestive heart failure
* No serious cardiac arrhythmias
* No evidence of recent prior myocardial infarction on EKG
* No clinical coronary artery disease

Pulmonary:

* No chronic obstructive pulmonary disease

Immunologic:

* No prior eczema
* HIV negative
* No immunocompromising conditions, (e.g., active autoimmune disease, leukemia, lymphoma, skin diseases, or open wounds)
* No clinical or laboratory evidence of an underlying immunosuppressive disorder
* No active or chronic infections
* No significant allergy or hypersensitivity to eggs

Other:

* No active seizure disorders
* No other malignancy within the past 2 years except stage I cervical cancer or basal cell skin cancer, provided the tumor has been successfully treated and patient is currently disease free
* No evidence of bone marrow toxicity
* No other concurrent medical illness that would preclude study
* No other contraindications to vaccinia virus administration
* No encephalitis
* Must be able to avoid close contact with children under 3 years of age; pregnant women; individuals with prior or active eczema or other open skin conditions; or immunosuppressed individuals for 7-10 days after each vaccination
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior vaccinia immunization required (e.g., smallpox vaccination)
* More than 8 weeks since prior immunotherapy and recovered
* No prior therapy with live vaccinia virus vector

Chemotherapy:

* More than 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior systemic corticosteroids
* No concurrent systemic corticosteroids
* No concurrent steroids

Radiotherapy:

* See Disease Characteristics
* More than 2 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* More than 4 weeks since prior surgery for primary tumor or metastatic lesions and recovered

Other:

* No concurrent immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. Kaufman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States